CLINICAL TRIAL: NCT04250376
Title: The Use of Transcranial Focused Ultrasound for the Treatment of Neurodegenerative Dementias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32222-1
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Parkinson Disease; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): All patients enrolled will receive transcranial focused ultrasound. Target location is dependent on patient condition.
  Interventions: Device: Focused Transcranial Ultrasound

INTERVENTIONS:
Device: Focused Transcranial Ultrasound — The FDA has determined the power intensity limits that are safe for clinical use; the proposed equipment works within these parameters. Furthermore, monitoring sessions up to one hour as proposed in this study are routinely used in patients even with acute brain injury at 2 megaHertz without any reports of complications induced by the ultrasound device. No brain heating, cavitation or bleeding has been identified with the proposed equipment and protocol. For each individual safety can be followed by performing a selective mental status exam at each session completion (for example for hippocampal targets, there will be a delayed recall memory test).

SUMMARY:
The purpose of this open label study is to evaluate longer term tolerability and early efficacy of transcranial ultrasound in the treatment of patients with mild cognitive impairment or dementia.

DETAILED DESCRIPTION:
The present study is designed as an open label study of patients with mild cognitive impairment (MCI) or dementia to evaluate longer term tolerability and early efficacy of transcranial ultrasound treatment.

Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures which are not affected by practice effects. For patients with amnestic predominant cognitive change, the target will be the mesial temporal lobe through a trans temporal scalp window. Targeting will include reference to scalp fiducials based on the obtained MRI and Transcranial Doppler (TCD) waveform confirmation will be obtained because of the ability of TCD to record Doppler signal from the posterior cerebral artery that runs medial to the mesial temporal lobe.

On the day of the ultrasound appointment, patients will undergo ten to thirty minutes of transcranial ultrasound treatment. The sonification device will be aimed at the hippocampus or the putamen and substantia nigra, depending on the predetermined condition. Targeting will include reference to scalp fiducials based on the obtained MRI; confirmation of target accuracy will either be obtained by Doppler waveform confirmation or optical tracking technology which co-registers patient neuroimaging with real space. Patients will undergo 8 total sessions of focused ultrasound. Patients will be evaluated at baseline and upon final ultrasound treatment using the same measures obtained upon entry. Safety and any adverse events will be monitored closely.

ELIGIBILITY:
Inclusion Criteria:

* CDR stage of at least 0.5 (mild cognitive impairment)
* At least one pathognomic imaging biomarker of a neurodegenerative process.

Exclusion Criteria:

* Cognitive decline clearly related to an acute illness
* Subjects unable to give informed consent
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
* Advanced terminal illness
* Advanced kidney, pulmonary, cardiac or liver failure
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Subjects with major depressive disorder
* Subjects with vascular causes of dementia

Ages: 45 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Quick Dementia Rating Scale | Baseline
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).

SECONDARY OUTCOMES:
Repeatable Battery Assessment for Neuropsychological Status (RBANS) | Baseline
  RBANS assesses immediate memory, visuospatial skill, language, attention, and delayed memory. Patient performance on each subscale immediate memory, language, attention, visuospatial, and delayed memory are scored relative to validated norms for same-aged peers. A change of 8+ points in the Total Scale score, 11+ points in the Immediate Memory score, 9+ points in the Language score, 4+ points on the Attention score, 14+ points is considered significant for the Visuospatial score, and 10+ points for the Delayed Memory score are considered significant.
Repeatable Battery Assessment for Neuropsychological Status (RBANS) | After final ultrasound (8 weeks from baseline)
  RBANS assesses immediate memory, visuospatial skill, language, attention, and delayed memory. Patient performance on each subscale immediate memory, language, attention, visuospatial, and delayed memory are scored relative to validated norms for same-aged peers. A change of 8+ points in the Total Scale score, 11+ points in the Immediate Memory score, 9+ points in the Language score, 4+ points on the Attention score, 14+ points is considered significant for the Visuospatial score, and 10+ points for the Delayed Memory score are considered significant.
Montreal Cognitive Assessment (MoCA) | Baseline
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
Montreal Cognitive Assessment (MoCA) | After final ultrasound (8 weeks from baseline)
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
Quick Dementia Rating Scale (QDRS) | After final ultrasound (8 weeks from baseline)
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon E Jordan, M.D., Principal Investigator — Neurology Management Associates
Locations (1):
- Neurological Associates of West LA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgess A, Dubey S, Yeung S, Hough O, Eterman N, Aubert I, Hynynen K. Alzheimer disease in a mouse model: MR imaging-guided focused ultrasound targeted to the hippocampus opens the blood-brain barrier and improves pathologic abnormalities and behavior. Radiology. 2014 Dec;273(3):736-45. doi: 10.1148/radiol.14140245. Epub 2014 Sep 15. PMID 25222068
- [Background] Chen K, Lu Z, Xin YC, Cai Y, Chen Y, Pan SM. Alpha-2 agonists for long-term sedation during mechanical ventilation in critically ill patients. Cochrane Database Syst Rev. 2015 Jan 6;1(1):CD010269. doi: 10.1002/14651858.CD010269.pub2. PMID 25879090
- [Background] Fitzgerald PJ. Is elevated norepinephrine an etiological factor in some cases of Alzheimer's disease? Curr Alzheimer Res. 2010 Sep;7(6):506-16. doi: 10.2174/156720510792231775. PMID 20626335
- [Background] Nir Y, Staba RJ, Andrillon T, Vyazovskiy VV, Cirelli C, Fried I, Tononi G. Regional slow waves and spindles in human sleep. Neuron. 2011 Apr 14;70(1):153-69. doi: 10.1016/j.neuron.2011.02.043. PMID 21482364
- [Background] Fucke T, Suchanek D, Nawrot MP, Seamari Y, Heck DH, Aertsen A, Boucsein C. Stereotypical spatiotemporal activity patterns during slow-wave activity in the neocortex. J Neurophysiol. 2011 Dec;106(6):3035-44. doi: 10.1152/jn.00811.2010. Epub 2011 Aug 17. PMID 21849616
- [Background] Iliff JJ, Goldman SA, Nedergaard M. Implications of the discovery of brain lymphatic pathways. Lancet Neurol. 2015 Oct;14(10):977-9. doi: 10.1016/S1474-4422(15)00221-5. No abstract available. PMID 26376966
- [Background] Jagust W. Is amyloid-beta harmful to the brain? Insights from human imaging studies. Brain. 2016 Jan;139(Pt 1):23-30. doi: 10.1093/brain/awv326. Epub 2015 Nov 27. PMID 26614753
- [Background] Jordao JF, Thevenot E, Markham-Coultes K, Scarcelli T, Weng YQ, Xhima K, O'Reilly M, Huang Y, McLaurin J, Hynynen K, Aubert I. Amyloid-beta plaque reduction, endogenous antibody delivery and glial activation by brain-targeted, transcranial focused ultrasound. Exp Neurol. 2013 Oct;248:16-29. doi: 10.1016/j.expneurol.2013.05.008. Epub 2013 May 21. PMID 23707300
- [Background] Kim H, Chiu A, Lee SD, Fischer K, Yoo SS. Focused ultrasound-mediated non-invasive brain stimulation: examination of sonication parameters. Brain Stimul. 2014 Sep-Oct;7(5):748-56. doi: 10.1016/j.brs.2014.06.011. Epub 2014 Jul 2. PMID 25088462
- [Background] Kress BT, Iliff JJ, Xia M, Wang M, Wei HS, Zeppenfeld D, Xie L, Kang H, Xu Q, Liew JA, Plog BA, Ding F, Deane R, Nedergaard M. Impairment of paravascular clearance pathways in the aging brain. Ann Neurol. 2014 Dec;76(6):845-61. doi: 10.1002/ana.24271. Epub 2014 Sep 26. PMID 25204284
- [Background] Lavialle M, Aumann G, Anlauf E, Prols F, Arpin M, Derouiche A. Structural plasticity of perisynaptic astrocyte processes involves ezrin and metabotropic glutamate receptors. Proc Natl Acad Sci U S A. 2011 Aug 2;108(31):12915-9. doi: 10.1073/pnas.1100957108. Epub 2011 Jul 13. PMID 21753079
- [Background] Lee W, Kim H, Jung Y, Song IU, Chung YA, Yoo SS. Image-guided transcranial focused ultrasound stimulates human primary somatosensory cortex. Sci Rep. 2015 Mar 4;5:8743. doi: 10.1038/srep08743. PMID 25735418
- [Background] Leinenga G, Gotz J. Scanning ultrasound removes amyloid-beta and restores memory in an Alzheimer's disease mouse model. Sci Transl Med. 2015 Mar 11;7(278):278ra33. doi: 10.1126/scitranslmed.aaa2512. PMID 25761889
- [Background] Leshchyns'ka I, Liew HT, Shepherd C, Halliday GM, Stevens CH, Ke YD, Ittner LM, Sytnyk V. Abeta-dependent reduction of NCAM2-mediated synaptic adhesion contributes to synapse loss in Alzheimer's disease. Nat Commun. 2015 Nov 27;6:8836. doi: 10.1038/ncomms9836. PMID 26611261
- [Background] Lim AS, Ellison BA, Wang JL, Yu L, Schneider JA, Buchman AS, Bennett DA, Saper CB. Sleep is related to neuron numbers in the ventrolateral preoptic/intermediate nucleus in older adults with and without Alzheimer's disease. Brain. 2014 Oct;137(Pt 10):2847-61. doi: 10.1093/brain/awu222. Epub 2014 Aug 20. PMID 25142380
- [Background] Lin GG, Scott JG. Investigations of the constitutive overexpression of CYP6D1 in the permethrin resistantLPR strain of house fly (Musca domestica). Pestic Biochem Physiol. 2011 Jun;100(2):130-134. doi: 10.1016/j.pestbp.2011.02.012. PMID 21765560
- [Background] Mander BA, Marks SM, Vogel JW, Rao V, Lu B, Saletin JM, Ancoli-Israel S, Jagust WJ, Walker MP. beta-amyloid disrupts human NREM slow waves and related hippocampus-dependent memory consolidation. Nat Neurosci. 2015 Jul;18(7):1051-7. doi: 10.1038/nn.4035. Epub 2015 Jun 1. PMID 26030850
- [Background] O'Donnell J, Ding F, Nedergaard M. Distinct functional states of astrocytes during sleep and wakefulness: Is norepinephrine the master regulator? Curr Sleep Med Rep. 2015 Mar;1(1):1-8. doi: 10.1007/s40675-014-0004-6. Epub 2015 Jan 29. PMID 26618103
- [Background] Ricci S, Dinia L, Del Sette M, Anzola P, Mazzoli T, Cenciarelli S, Gandolfo C. Sonothrombolysis for acute ischaemic stroke. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD008348. doi: 10.1002/14651858.CD008348.pub2. PMID 22696378
- [Background] Scarcelli T, Jordao JF, O'Reilly MA, Ellens N, Hynynen K, Aubert I. Stimulation of hippocampal neurogenesis by transcranial focused ultrasound and microbubbles in adult mice. Brain Stimul. 2014 Mar-Apr;7(2):304-7. doi: 10.1016/j.brs.2013.12.012. Epub 2014 Jan 28. PMID 24629831
- [Background] Schlesinger D, Benedict S, Diederich C, Gedroyc W, Klibanov A, Larner J. MR-guided focused ultrasound surgery, present and future. Med Phys. 2013 Aug;40(8):080901. doi: 10.1118/1.4811136. PMID 23927296
- [Background] Seitz DP, Reimer CL, Siddiqui N. A review of epidemiological evidence for general anesthesia as a risk factor for Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Dec 2;47:122-7. doi: 10.1016/j.pnpbp.2012.06.022. Epub 2012 Jul 4. PMID 22771690
- [Background] Sevigny J, Chiao P, Bussiere T, Weinreb PH, Williams L, Maier M, Dunstan R, Salloway S, Chen T, Ling Y, O'Gorman J, Qian F, Arastu M, Li M, Chollate S, Brennan MS, Quintero-Monzon O, Scannevin RH, Arnold HM, Engber T, Rhodes K, Ferrero J, Hang Y, Mikulskis A, Grimm J, Hock C, Nitsch RM, Sandrock A. The antibody aducanumab reduces Abeta plaques in Alzheimer's disease. Nature. 2016 Sep 1;537(7618):50-6. doi: 10.1038/nature19323. PMID 27582220
- [Background] Shteamer JW, Dedhia RC. Sedative choice in drug-induced sleep endoscopy: A neuropharmacology-based review. Laryngoscope. 2017 Jan;127(1):273-279. doi: 10.1002/lary.26132. Epub 2016 Jul 1. PMID 27363604
- [Background] Siemers ER, Sundell KL, Carlson C, Case M, Sethuraman G, Liu-Seifert H, Dowsett SA, Pontecorvo MJ, Dean RA, Demattos R. Phase 3 solanezumab trials: Secondary outcomes in mild Alzheimer's disease patients. Alzheimers Dement. 2016 Feb;12(2):110-120. doi: 10.1016/j.jalz.2015.06.1893. Epub 2015 Aug 1. PMID 26238576
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Thal DR, Walter J, Saido TC, Fandrich M. Neuropathology and biochemistry of Abeta and its aggregates in Alzheimer's disease. Acta Neuropathol. 2015 Feb;129(2):167-82. doi: 10.1007/s00401-014-1375-y. Epub 2014 Dec 23. PMID 25534025
- [Background] Whittington RA, Bretteville A, Dickler MF, Planel E. Anesthesia and tau pathology. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Dec 2;47:147-55. doi: 10.1016/j.pnpbp.2013.03.004. Epub 2013 Mar 25. PMID 23535147
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Svetoni F, Frisone P, Paronetto MP. Role of FET proteins in neurodegenerative disorders. RNA Biol. 2016 Nov;13(11):1089-1102. doi: 10.1080/15476286.2016.1211225. Epub 2016 Jul 14. PMID 27415968
- [Background] Bohnen NI, Albin RL, Koeppe RA, Wernette KA, Kilbourn MR, Minoshima S, Frey KA. Positron emission tomography of monoaminergic vesicular binding in aging and Parkinson disease. J Cereb Blood Flow Metab. 2006 Sep;26(9):1198-212. doi: 10.1038/sj.jcbfm.9600276. Epub 2006 Jan 18. PMID 16421508
- [Background] Kotagal V, Bohnen NI, Muller ML, Frey KA, Albin RL. Cerebral Amyloid Burden and Hoehn and Yahr Stage 3 Scoring in Parkinson Disease. J Parkinsons Dis. 2017;7(1):143-147. doi: 10.3233/JPD-160985. PMID 28106566
- [Background] Shah N, Frey KA, Muller ML, Petrou M, Kotagal V, Koeppe RA, Scott PJ, Albin RL, Bohnen NI. Striatal and Cortical beta-Amyloidopathy and Cognition in Parkinson's Disease. Mov Disord. 2016 Jan;31(1):111-7. doi: 10.1002/mds.26369. Epub 2015 Sep 18. PMID 26380951
- [Background] Hsiao IT, Weng YH, Hsieh CJ, Lin WY, Wey SP, Kung MP, Yen TC, Lu CS, Lin KJ. Correlation of Parkinson disease severity and 18F-DTBZ positron emission tomography. JAMA Neurol. 2014 Jun;71(6):758-66. doi: 10.1001/jamaneurol.2014.290. PMID 24756323
- [Background] Petrou M, Bohnen NI, Muller ML, Koeppe RA, Albin RL, Frey KA. Abeta-amyloid deposition in patients with Parkinson disease at risk for development of dementia. Neurology. 2012 Sep 11;79(11):1161-7. doi: 10.1212/WNL.0b013e3182698d4a. Epub 2012 Aug 29. PMID 22933741
- [Background] Edison P, Rowe CC, Rinne JO, Ng S, Ahmed I, Kemppainen N, Villemagne VL, O'Keefe G, Nagren K, Chaudhury KR, Masters CL, Brooks DJ. Amyloid load in Parkinson's disease dementia and Lewy body dementia measured with [11C]PIB positron emission tomography. J Neurol Neurosurg Psychiatry. 2008 Dec;79(12):1331-8. doi: 10.1136/jnnp.2007.127878. Epub 2008 Jul 24. PMID 18653550
- [Background] Gomperts SN, Rentz DM, Moran E, Becker JA, Locascio JJ, Klunk WE, Mathis CA, Elmaleh DR, Shoup T, Fischman AJ, Hyman BT, Growdon JH, Johnson KA. Imaging amyloid deposition in Lewy body diseases. Neurology. 2008 Sep 16;71(12):903-10. doi: 10.1212/01.wnl.0000326146.60732.d6. PMID 18794492
- [Background] Burack MA, Hartlein J, Flores HP, Taylor-Reinwald L, Perlmutter JS, Cairns NJ. In vivo amyloid imaging in autopsy-confirmed Parkinson disease with dementia. Neurology. 2010 Jan 5;74(1):77-84. doi: 10.1212/WNL.0b013e3181c7da8e. PMID 20038776
- [Background] Ito H, Shinotoh H, Shimada H, Miyoshi M, Yanai K, Okamura N, Takano H, Takahashi H, Arakawa R, Kodaka F, Ono M, Eguchi Y, Higuchi M, Fukumura T, Suhara T. Imaging of amyloid deposition in human brain using positron emission tomography and [18F]FACT: comparison with [11C]PIB. Eur J Nucl Med Mol Imaging. 2014 Apr;41(4):745-54. doi: 10.1007/s00259-013-2620-7. PMID 24233004
- [Background] Sivanesam K, Andersen NH. Modulating the Amyloidogenesis of alpha-Synuclein. Curr Neuropharmacol. 2016;14(3):226-37. doi: 10.2174/1570159x13666151030103153. PMID 26517049
- [Background] Terrelonge M Jr, Marder KS, Weintraub D, Alcalay RN. CSF beta-Amyloid 1-42 Predicts Progression to Cognitive Impairment in Newly Diagnosed Parkinson Disease. J Mol Neurosci. 2016 Jan;58(1):88-92. doi: 10.1007/s12031-015-0647-x. Epub 2015 Sep 2. PMID 26330275
- [Background] Stav AL, Aarsland D, Johansen KK, Hessen E, Auning E, Fladby T. Amyloid-beta and alpha-synuclein cerebrospinal fluid biomarkers and cognition in early Parkinson's disease. Parkinsonism Relat Disord. 2015 Jul;21(7):758-64. doi: 10.1016/j.parkreldis.2015.04.027. Epub 2015 May 2. PMID 25971633
- [Background] Petrou M, Dwamena BA, Foerster BR, MacEachern MP, Bohnen NI, Muller ML, Albin RL, Frey KA. Amyloid deposition in Parkinson's disease and cognitive impairment: a systematic review. Mov Disord. 2015 Jun;30(7):928-35. doi: 10.1002/mds.26191. Epub 2015 Apr 16. PMID 25879534
- [Background] Walker L, McAleese KE, Thomas AJ, Johnson M, Martin-Ruiz C, Parker C, Colloby SJ, Jellinger K, Attems J. Neuropathologically mixed Alzheimer's and Lewy body disease: burden of pathological protein aggregates differs between clinical phenotypes. Acta Neuropathol. 2015 May;129(5):729-48. doi: 10.1007/s00401-015-1406-3. Epub 2015 Mar 11. PMID 25758940